CLINICAL TRIAL: NCT05842681
Title: Role of Add-on Azithromycin in the Management of Patients With Acute Exacerbation of Idiopathic Pulmonary Fibrosis
Brief Title: Azithromycin in the Management of Patients With Acute Exacerbation of Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Shaddad, Lecturer of pulmonary medicine Assuit university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2516771716
Record Dates: First submitted 2023-04-23; First posted 2023-05-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Azithromycin; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional therapy group (Active Comparator): Patients will receive conventional treatment for acute exacerbation of IPF, including pulse corticosteroid therapy and supportive treatment, and oxygen therapy.
  Interventions: Drug: Methylprednisolone
- Add-on Azithromycin (Active Comparator): Patients will receive conventional therapy and Add-on Azithromycin 500 mg single daily dose for five days
  Interventions: Drug: Azithromycin; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Azithromycin — A single daily oral dose of Azithromycin tablet 500 mg for five days
  Other Names: azithromycin 500 mg oral tablet
  Arms: Add-on Azithromycin
Drug: Methylprednisolone — methylprednisolone 500 mg single intra-venous daily dose for three days
  Other Names: methylprednisolone 500 mg

SUMMARY:
This randomized controlled trial evaluates the therapeutic role of azithromycin in acute exacerbations of idiopathic pulmonary fibrosis (AE-IPF). Baseline severity classification and stratification were performed using the SCALE-IPF framework (Severity Classification and Lung Evaluation for Prognosis in IPF; locked April 2023) to ensure balanced disease severity across randomized arms. End-of-study analyses included descriptive and stratified phenotyping using the IPIM (Idiopathic Pulmonary Fibrosis Phenotypes Identification Model; locked April 2023).

Both frameworks were developed within the Assiut University IPF Research Program (2022-2026), a coordinated institutional effort investigating clinical, prognostic, and therapeutic dimensions of IPF. Neither framework altered randomization procedures, treatment allocation, or study endpoints; they were applied to improve standardization, reproducibility, and interpretability of results.

DETAILED DESCRIPTION:
This randomized, open-label controlled trial forms part of the Assiut University IPF Research Program (2022-2026). An initial target of 130 patients with clinically mild or early-moderate acute exacerbation of idiopathic pulmonary fibrosis (AE-IPF) was specified for enrollment and randomized to receive standard therapy with or without azithromycin.

SCALE-IPF (Severity Classification and Lung Evaluation for Prognosis in IPF; locked April 2023, archived November 2025, digital object identifier [DOI] 10.5281/zenodo.17575973) served as the prespecified baseline severity classification and stratification framework. IPIM (Idiopathic Pulmonary Fibrosis Phenotypes Identification Model; locked April 2023, archived November 2025, DOI 10.5281/zenodo.17576160) was applied as a predefined phenotypic framework integrating clinical, functional, and radiological domains.

Severity and phenotypic frameworks were used exclusively to define eligibility and baseline characterization. They did not influence randomization procedures, treatment allocation, trial conduct, or study endpoints, and were applied to support reproducibility and structured interpretation of therapeutic effects across severity and phenotypic spectra.

ELIGIBILITY:
Inclusion Criteria:

* Baseline disease severity classified as mild or early-moderate according to the SCALE-IPF (locked April 2023) threshold ≤ 13 points.
* Participation within the Assiut University IPF Research Program (2022-2026).

Exclusion Criteria:

* Age: less than 18 years.
* Patients with any severity other than mild or early-moderate acute exacerbation of IPF according to SCALE-IPF (locked April 2023).
* Patients with multislice computed tomography with a radiological pattern rather than usual interstitial pneumonitis (UIP).
* Unstable patients need mechanical ventilation or Respiratory Intensive Care Unit admission.
* Patients with end-organ failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Hospital stay | 5-10 Days ( Days of Hospital admission until improvement and discharge)
  the main aime of the study to assess the hospital stay expressed in days in the Add-on Azithromycin 500 mg single oral daily dose in comparison to the conventional therapy group only

SECONDARY OUTCOMES:
Change in clinical outcome measures stratified by SCALE-IPF severity | From randomization (Day 1) to Month 3 post-enrollment.
  Evaluate the treatment response and short-term progression of AE-IPF patients across baseline severity strata as defined by the SCALE-IPF classification (locked April 2023).
  Outcomes include improvement in oxygenation, radiological resolution, and need for hospitalization.
  This will assess whether baseline SCALE-IPF strata correlate with therapeutic response and clinical stability.
Association between SCALE-IPF severity and one-year mortality | Baseline to 12 months post-randomization.
  Determine whether baseline SCALE-IPF severity independently predicts 12-month all-cause mortality following acute exacerbation in both treatment arms.
  This analysis provides validation of the SCALE-IPF prognostic gradient within a randomized framework.
Correlation between azithromycin response and IPIM phenotypic clusters | Baseline to 12 months post-randomization.
  Analysis comparing treatment outcomes across IPIM-defined phenotypic clusters
Event-free survival across SCALE-IPF strata | Baseline to 12 months post-randomization.
  Compare event-free survival (freedom from recurrent AE, hospitalization, or death) between azithromycin and control groups across SCALE-defined severity categories.

OTHER OUTCOMES:
Analytical validation of SCALE-IPF and IPIM within the randomized AE-IPF cohort | Baseline to 12 months post-randomization.
  Evaluate the performance, calibration, and clinical concordance of the two institutional frameworks-SCALE-IPF (randomization classifier) and IPIM (descriptive phenotype model)-within the azithromycin randomized trial population.

CONTACTS AND LOCATIONS:
Overall Officials: ahmad M shaddad, Principal Investigator — Assiut university-Faculty of Medicine
Locations (2):
- Egypt (2):
  - Assiut university-Faculty of Medicine, Asyut
  - Faculty of Medicine Assuit University, Asyut

IPD SHARING:
Plan to Share IPD: No